CLINICAL TRIAL: NCT03081936
Title: Comparative Effects of A1 Versus A2®Cow Milk Based Formula and Breast Feeding on Alimentation and Gastrointestinal Digestion for the Infant: a Pilot Double-blinded, Randomized, Controlled Parallel Study
Brief Title: Comparative A1 vs A2 Formula and Breast Feeding on Alimentation and Gastrointestinal Digestion for the Infant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: a2 Milk Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 15-SC-6-A2-003
Record Dates: First submitted 2016-11-01; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Intestinal Absorption
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A1 formula (Active Comparator): Oral consumption of Nutricia Aptamil Stage 1 formula (traditional cow milk)
  Interventions: Dietary Supplement: Oral consumption of Nutricia Aptamil Stage 1 formula
- A2 formula (Experimental): Oral consumption of a2® Platinum Stage 1 formula (containing 100% A2® beta -casein)
  Interventions: Dietary Supplement: Oral consumption of a2® Platinum Stage 1 formula
- Breast feeding (Active Comparator): Oral consumption of breast milk
  Interventions: Dietary Supplement: Oral consumption of breast milk

INTERVENTIONS:
Dietary Supplement: Oral consumption of Nutricia Aptamil Stage 1 formula — Daily oral consumption of Nutricia Aptamil Stage 1 formula
  Arms: A1 formula
Dietary Supplement: Oral consumption of a2® Platinum Stage 1 formula — Daily oral consumption of a2® Platinum Stage 1 formula
  Arms: A2 formula
Dietary Supplement: Oral consumption of breast milk — Daily oral consumption of breast milk
  Arms: Breast feeding

SUMMARY:
This pilot study primarily aimed to compare effects of breast feeding, A1 versus A2®cow milk based formula on alimentation and gastrointestinal digestion. The impact of the study products on fecal myeloperoxidase (MPO), short-chain fatty acid (SCFA), secretory immunoglobulin A (sIgA) concentration, gastrointestinal tolerance, defecating habit and infant growth were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Willing to formula feeding and consume 600ml or more of IF each day;
* Have normal electrocardiograms (ECG) and blood pressure during quiet respiration.
* Agree not to take any medication, supplements, nutrition or other dairy products including acidophilus milk;
* Parent(s) or legal guardian's consent to the study and willing to comply with study procedures;
* Parent(s) or guardian of infant agrees not to enroll infant another clinical study while participating in this study;
* Fully understand the nature, objective, benefit and the potential risks and side effects of the study.

Exclusion Criteria:

* Twins, multiple birth, low birth weight children, over birth weight children or early birth children with gestational age less than 37 weeks;
* During pregnancy, the mothers had pregnancy complications or other disease that may affect the results;
* Having serious diseases that may affect study interventions, such as neonatal sepsis, pneumonia (associated with respiratory failure), heart failure and other disease;
* Having neonatal diarrhea or acute respiratory infections within 48hours before enrollment;
* Having potential metabolic diseases, chronic diseases, congenital malformations, central nervous system disorders, neuromuscular disorders or diseases affecting bone metabolism that may affect growth or the study results;
* Having taken any food containing prebiotics or probiotics tithing 15 days of enrollment;
* Body weight-to-height Z-value <-3 according to the standard of the World Health Organization (WHO);
* Receiving hormone therapy and intravenous nutrition;
* Lactose intolerance or allergic to ingredients of study product;
* Have history of faecal impaction;
* Have participated in similar dairy or probiotics-containing product's clinical trials within 3 months before the screening;
* Currently taking medicines for cardiovascular or metabolic disease ;
* Currently suffering from any gastrointestinal disorders or gastrointestinal disease , including but not limited to: irritable bowel syndrome, colitis, ulcerative colitis, celiac disease, irritable bowel syndrome(IBS);
* Had hospitalizations within 3 months before screening;
* According to investigator's judgment, current frequent users of drugs which may affect the gastrointestinal function or immune system;
* Unable to comply the study schedule.

Ages: 40 Days to 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Stool frequency | Baseline, Week 8
  Change from Baseline weekly average of the number of defecation per day at 8 weeks

SECONDARY OUTCOMES:
Stool consistency | Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8
  Weekly average score of stool consistency
Stool color | Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8
  Weekly average score of stool color
Fecal Myeloperoxidase (MPO) concentration | Baseline, Day 7, Day 56
Fecal Short Chain Fatty Acid (SCFA) concentration | Baseline, Day 7, Day 56
  Acetic Acid , Propanoic Acid, Butanoic Acid, Total SCFA
Fecal sIgA concentration | Baseline, Day 7, Day 56
Fecal microflora counts | Baseline, Day 7, Day 56
  Bifidobacterium, Lactobacillus, Clostridium perfringens
Body weight | Baseline, Day 7, Day 56
  Body weight (unit: g)
Body height | Baseline, Day 7, Day 56
  Body height (unit: cm)
Head circumstance | Baseline, Day 7, Day 56
  Head circumstance (unit: cm)
Chest circumstance | Baseline, Day 7, Day 56
  Chest circumstance (unit: cm)
Cry frequency | Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8
  Weekly average of cry frequency per day
Cry duration | Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8
  Weekly average of cumulative cry duration per day
Sleep duration | Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8
  Weekly average of cumulative sleep duration per day
Milk regurgitation frequency | Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8
  Weekly average of milk regurgitation frequency per day

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Zhang, MD, Study Director — Sprim (Shanghai) Consulting Co., Ltd.

IPD SHARING:
Plan to Share IPD: No